CLINICAL TRIAL: NCT01654588
Title: Different End Points for Bronchial Hyperactivity (BHR) Tests, What Comes First?
Brief Title: Different End Points for Bronchial Hyperactivity (BHR) Tests.
Status: Completed | Type: Observational
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Avigdor Mandelberg, Director, Pediatric Pulmonry Unit, Wolfson Medical Center
Other Study IDs: AD-S
Record Dates: First submitted 2011-07-26; First posted 2012-08-01 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Bronchial Hyperreactivity
Keywords: BRONCHIAL CHALLANGE TEST, ASTHMA, METACHLINE, ADENOSINE
MeSH Terms: conditions — Bronchial Hyperreactivity; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Bronchial challenge tests (BCT) are being used to diagnose bronchial hyperactivity (BHR) and quantify its severity.In older children and adults, BCT is done using spirometry to measure the value of 20% fall in FEV1 as an indicator for positive reactivity.

However, in young children and infants that cannot perform spirometry, other measurements are used as indicators for BHR. Traditionally, in these populations, appearance of wheezing on auscultation is used as the indicator for BHR. More recently, other measures like 50% increase in respiratory rate or 5% decreases in oxygen saturation are mentioned as possible options to determine positive BHR. Nevertheless, as these measurements probably measure different parameters they could vary in time of appearance.

The investigators also noted that in older children who perform spirometry, the order of appearance of these different physiologic measures is not constant.

Decrease in O2 saturation, appearance of wheezing and increase in respiratory rate (RR) do not all appear at the same time and not in the same order of events.

Some children are noted to have a decrease in FEV1 without wheezing - those children can be difficult to diagnose as asthmatics in the primary care setting where asthma is being diagnosed on clinical grounds alone: wheezing and response to bronchodilators. Children who do not wheeze are difficult to diagnose and therefore, are not getting the appropriate treatment.

Nevertheless, the data in current literature is very scant or not existing regarding these issues. Thus the investigators designed a study to prospectively try to answer the questions: do clinically significant differences exist in the concentration of the metacholine and / or adenosine at the time time of appearances of these parameters, what comes first, and if so, how does it affect the diagnosis and the severity assessment of HRA in different age groups?

DETAILED DESCRIPTION:
Bronchial challenge tests (BCT) are being used to diagnose bronchial hyperactivity (BHR) and quantify its severity.

In older children and adults, BCT is done using spirometry to measure the value of 20% fall in FEV1 as an indicator for positive reactivity. However, in young children and infants that cannot perform spirometry, other measurements are used as indicators for BHR. Traditionally, in these populations, appearance of wheezing on auscultation is used as the indicator for BHR. More recently, other measures like 50% increase in respiratory rate or 5% decreases in oxygen saturation are mentioned as possible options to determine positive BHR. Nevertheless, as these measurements probably measure different parameters they could vary in time of appearance.

The investigators also noted that in older children who perform spirometry, the order of appearance of these different physiologic measures is not constant.

Decrease in O2 saturation, appearance of wheezing and increase in respiratory rate (RR) do not all appear at the same time and not in the same order of events.

Some children are noted to have a decrease in FEV1 without wheezing - those children can be difficult to diagnose as asthmatics in the primary care setting where asthma is being diagnosed on clinical grounds alone: wheezing and response to bronchodilators. Children who do not wheeze are difficult to diagnose and therefore, are not getting the appropriate treatment.

Nevertheless, the data in current literature is very scant or not existing regarding these issues. Thus the investigators designed a study to prospectively try to answer the questions: do clinically significant differences exist in the time of appearances of these parameters and if so, how does it affect the diagnosis and the severity assessment of HRA in different age groups? in this study we measure the metacholine and / or adenosine concentration at the time when the following parameters appear (what comes first): 20% fall in FEV1, 5% fall in oxygen saturation, 50% rise in respiratory rate, wheezing heard by the investigators using stethoscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for HRA trigger testing

Exclusion Criteria:

* None

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients referred for HRA trigger testing.
Sampling Method: Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Which of the outcome ends points measures comes first in the diagnosis of bronchial hypersensitiveness. | On which metacholine and / or adenosine increasing concentrations, there are 20% fall in FEV1 and / or 5% decrease in saturation and / or 50% increase in RR. Which comes first. Time frame: each BHR tests last up to two hours.
  Increasing concentrations of Metacholine or adenosine inhalations are given until there are 20% fall in FEV1 and / or 5% decrease in saturation and / or 50% increase in RR. The concentrations on which these outcomes occur are measured.

SECONDARY OUTCOMES:
Age influence on which comes first outcomes. | The time frame of the study: four years.
  Age in years and months will be recorded. Age influence on the distribution of the main outcome - which comes first - will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Avigdor Madnelberg, MD, Principal Investigator — The Sackler School of Medicine, Tel-Aviv University, Israel; Avigdor Mandelberg, MD, Principal Investigator — Tha Sackler School of Medicine, Tel-Aviv University, Israel
Locations (1):
- The Edith Wlofson Medical Center, Holon, Israel

REFERENCES:
- [Derived] Ater D, Amirav I, Attias M, Nakash E, Newhouse MT, Mandelberg A. Evaluation of clinically and physiologically atypical asthma: If it doesn't wheeze it may still be asthma. J Asthma. 2019 Jan;56(1):21-26. doi: 10.1080/02770903.2018.1424194. Epub 2018 Feb 2. PMID 29393720